CLINICAL TRIAL: NCT02588157
Title: Videolaryngoscopes for Rapid Sequence Intubation
Brief Title: Effect of Cricoid Pressure on Macintosh, McGrath X-Blade and Glidescope Videolaryngoscopes in Rapid Sequence Induction Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: KOÜ KAEK 2015/267
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Rapid Sequence Induction Intubation
Keywords: Rapid sequence induction intubation; McGrath X-Blade; Glidescope; Macintosh

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- İnsertion time (Active Comparator): handling the device till the glottic visualisation of Macintosh, McGrath MAC X-Blade and Glidescope
  Interventions: Device: Macintosh; Device: Glidescope; Device: McGrath MAC X-Blade
- intubation time (Active Comparator): handling the device till seeing the endotracheal tube entering from the vocal cords Macintosh, McGrath MAC X-Blade and Glidescope
  Interventions: Device: Macintosh; Device: Glidescope; Device: McGrath MAC X-Blade

INTERVENTIONS:
Device: Macintosh — Direct laryngoscopy
  Other Names: direct laryngoscopy
Device: Glidescope — Glidescope videolaryngoscope
  Other Names: videolaryngoscope
Device: McGrath MAC X-Blade — McGrath MAC X-Blade videolaryngoscope
  Other Names: videolaryngoscope

SUMMARY:
Non- Fasted patients need rapid sequence intubation. The investigators aimed to compare the intubation times of Macintosh , and McGrath X-Blade or Glidescope in these Ascenario.

DETAILED DESCRIPTION:
The investigators fecidedir to enroll the ASA I-II 120 patients and divided them into three groups ( Macintosh / McGarth X-Blade / Glidescope). The investigators recorded the patients' airway data and demographic variables. All patients were premeditated with midazolam. Standard monitoring including electrocardiogram, non invasive blood pressure, pulse oximetry, heart rate were recorded before induction , after induction, after the device insertion and every 1 minutes after intubation. Cormac-Lehan grades with these video laryngoscope were recorded also. We recorded the optimization maneuvers ( like handling force, reinserting, cricoid pressure). Bloodstaining on the devices after removal were recorded as mucosal damage. Teeth, tongue, lip damage were also recorded. Sore throat, bronchospasm, wheezing were recored at recovery unit.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* BMI< 30
* 18-65 years of age

Exclusion Criteria:

* known difficult airway
* BMI > 30
* < 18 years of age
* > 65 years of age
* known respiratory tract infection in 10 days
* pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
cormack lehane grade with cricoid pressure | 1 minutes
intubation time | 2 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)